CLINICAL TRIAL: NCT05606991
Title: The Impact of 2 Weeks CPAP Withdrawal on Brain Waste Clearance in Adults With Severe Obstructive Sleep Apnoea - A Randomised Controlled Crossover Trial
Brief Title: The Effect of OSA on Brain Waste Clearance
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Woolcock Institute of Medical Research (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BrainOSA-0522
Record Dates: First submitted 2022-07-12; First posted 2022-11-07 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Obstructive Sleep Apnea; Dementia; Cognitive Impairment
Keywords: Obstructive sleep apnea; Brain waste clearance; Glymphatic system; Continuous positive airway pressure therapy; CPAP; Dementia; Cognitive impairment
MeSH Terms: conditions — Sleep Apnea, Obstructive; Dementia; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomized controlled crossover trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP on (No Intervention): Participants will continue with their usual continuous positive airway pressure (CPAP) therapy as advised by their treating physician.
- CPAP off (Experimental): Participants will be weaned off their usual continuous positive airway pressure (CPAP) therapy and enter a 2-week period of non-treatment.
  Interventions: Other: CPAP Withdrawal

INTERVENTIONS:
Other: CPAP Withdrawal — Complete withdrawal of continuous positive airway pressure (CPAP) therapy for a 2-week period.
  Arms: CPAP off

SUMMARY:
Recent ground-breaking research has shown that clearance of toxic neuro-metabolites from the brain including the proteins β-Amyloid (Aβ) and tau that form dementia causing plaques and tangles is markedly impaired when sleep is disturbed. This suggests that dementia risk may be increased in people with sleep disorders such as obstructive sleep apnea (OSA). Longitudinal studies have linked OSA with a 70-85% increased risk for mild cognitive impairment and dementia.

Despite this strong link, little is known about the OSA-specific mechanistic underpinnings. It is not fully understood as to how sleep disturbance in OSA inhibit brain glymphatic clearance. However, it is known that OSA inhibits slow wave sleep, profoundly activates sympathetic activity, and elevates blood pressure - particularly during sleep. These disturbances have, in turn, been shown to independently inhibit glymphatic function. Previous studies have attempted to sample human cerebrospinal fluid (CSF) involved in glymphatic clearance for dementia biomarkers during sleep. However, these studies were severely limited by the need for invasive CSF sampling. To address this problem, a set of newly available, highly sensitive blood based SIMOA assays will be used to study glymphatic function in people treated for severe OSA who undergo CPAP withdrawal. Furthermore, novel methods will be utilized to capture changes in slow wave sleep, blood pressure and brain blood flow together with sleep-wake changes in blood levels of excreted neuro-metabolites to define the pathophysiological mechanisms that inhibit brain cleaning in OSA.

DETAILED DESCRIPTION:
Dementia is a neurodegenerative disease characterized by cognitive dysfunction affecting aspects of memory and learning. Although the mechanisms that underlie the pathophysiology of dementia are still unclear, in the past decade there has been a focus on the adverse impact of sleep disturbance on brain waste disposal via the glymphatic system. The glymphatic system is a recently discovered brain-wide perivascular passageway that transports toxic neuro-metabolites (e.g.: amyloid beta, or Aβ) out of the brain to the blood via the cerebrospinal fluid. Newer research has shown that the glymphatic system becomes particularly active during sleep, clearing metabolites twice as fast compared with wakefulness. Obstructive sleep apnea (OSA), a sleep disorder characterized by periods of intermittent hypoxia and sleep fragmentation due to obstructed breathing, has traditionally been causatively linked to the development of hypertension and cognitive dysfunction. Further to this, recent epidemiological studies have also linked OSA to an increased risk for both dementia and its prodromal state - mild cognitive impairment. There is emerging evidence to suggest that OSA might chronically impair glymphatic clearance of Aβ42 from the brain and facilitate the formation of Aβ plaques that characterize Alzheimer's Disease.

Recent ground-breaking research has shown that clearance of toxic neuro-metabolites from the brain including the proteins Aβ and tau that form dementia causing plaques and tangles is markedly impaired when sleep is disturbed. This suggests that dementia risk may be increased in people with sleep disorders such as OSA. Longitudinal studies have linked OSA with a 70-85% increased risk for mild cognitive impairment and dementia.

Despite this strong link, little is known about the OSA-specific mechanistic underpinnings. It is not fully understood as to how sleep disturbance in OSA inhibit brain glymphatic clearance. However, it is known that OSA inhibits slow wave sleep, profoundly activates sympathetic activity, and elevates blood pressure - particularly during sleep. These disturbances have, in turn, been shown to independently inhibit glymphatic function. Previous studies have attempted to sample human cerebrospinal fluid (CSF) involved in glymphatic clearance for dementia biomarkers during sleep. However, these studies were severely limited by the need for invasive CSF sampling. To address this problem, this proposed study will use a set of newly available, highly sensitive blood based SIMOA assays to study glymphatic function in people treated for severe OSA who undergo CPAP withdrawal. Furthermore, novel methods will be utilized to capture changes in slow wave sleep, blood pressure and brain blood flow together with sleep-wake changes in blood levels of excreted neuro-metabolites to define the pathophysiological mechanisms that inhibit brain cleaning in OSA.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling adults aged 35-65 years.
* Polysomnography-confirmed severe OSA with apnea hypopnea index (AHI) ≥ 30/hour, with Non-Rapid Eye Movement (NREM) AHI ≥ 15/hour.
* Established CPAP use for treatment of OSA with compliance of > 3 months, with ≥ 5 hours use per night for > 5 nights per week.
* Willing to withdraw from CPAP use for 14 nights.
* Able to give informed verbal and written consent.
* Fluent in spoken, and comprehension of English.

Exclusion Criteria:

* Commercial drivers (e.g.: drivers of heavy vehicles, public passenger vehicles, or vehicles requiring dangerous goods driver license).
* History of severe cardiovascular disease (e.g.: stroke, myocardial infarction, atrial fibrillation).
* Presence of cognitive impairment and/or established diagnosis of dementia.
* Regular use of medications which affect sleep (e.g.: benzodiazepines, opioids, stimulants, sedating antihistamines).
* Regular 24-hour shift workers, presence of jetlag, or history of trans-meridian travel (crossing 2 or more time zones) in the past 2 weeks.
* Advice against withdrawal of CPAP treatment, as determined by the participant's treating physician or study physician.
* Vulnerable to driving impairment without CPAP therapy/upon withdrawal of CPAP therapy, as assessed by: (a) positive response(s) to screening questions in the modified ASTN-Motor Vehicle Accident Questionnaire, reporting driving accidents and/or impairments prior to established CPAP therapy; AND/OR (b) the participant's treating physician.
* Prior history of severe COVID-19 infection involving significant neurological symptoms (e.g.: reduced level of consciousness, delirium, encephalopathy) - warranting hospitalization.
* Current COVID-19 infection and/or experience of ongoing symptoms/sequelae following a recent COVID-19 infection.
* Not up to date with the COVID-19 vaccination schedule - as per the current Australian Technical Advisory Group on Immunization (ATAGI) definition for individuals aged 16 years and over - at the time of writing this Protocol, defined as having:

  1. Received 2 primary doses of any Therapeutic Goods Administration (TGA)-approved or TGA-recognized COVID-19 vaccine at least 14 days apart (except for the Janssen COVID-19 vaccine, where only 1 primary dose is required); PLUS
  2. A booster dose of a TGA-approved COVID-19 vaccine (Pfizer, Moderna or AstraZeneca) at a recommended interval of 3-6 months after the receipt of 2nd primary dose; OR
  3. For severely immunocompromised individuals: received 3 primary doses of any TGA-approved or TGA-recognized COVID-19 vaccine, with dose 3 administered within 6 months of receiving dose 2.
* Other medical conditions deemed by study physicians to warrant exclusion.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Changes in sleep-wake amplitudes (peak-trough) of blood levels of Aβ | Pre- and 2 weeks post-intervention
  Difference between the CPAP on and CPAP off conditions in sleep-wake amplitudes (peak-trough) of blood levels of Aβ (Aβ40/Aβ42 ratio), as measured by SIMOA blood neuro-metabolite assays.

SECONDARY OUTCOMES:
Changes in NREM slow wave parietal cortex activity | Pre- and 2 weeks post-intervention
  Differences between the CPAP on and CPAP off conditions in NREM slow wave parietal cortex activity as measured by high-density EEG (HD-EEG).
Changes in brain tissue oxygenation during sleep | Pre- and 2 weeks post-intervention
  Differences between the CPAP on and CPAP off conditions in brain tissue oxygenation, as measured by oxygenated and deoxygenated hemoglobin using functional Near Infrared Spectroscopy (fNIRS).
Changes in brain blood volume during sleep | Pre- and 2 weeks post-intervention
  Differences between the CPAP on and CPAP off conditions in brain blood volume during sleep, estimated by changes in total hemoglobin using functional Near Infrared Spectroscopy (fNIRS).
Changes in sympathetic and parasympathetic activity during wake and sleep periods | Pre- and 2 weeks post-intervention
  Differences between the CPAP on and CPAP off conditions in sympathetic and parasympathetic activity during wake and sleep periods, as measured by heart rate variability (HRV) analysis of electrocardiogram (ECG) readings.
Changes in sleep-wake amplitudes (peak-trough) of blood levels of p-tau-217 | Pre- and 2 weeks post-intervention
  Difference between the CPAP on and CPAP off conditions in sleep-wake amplitudes (peak-trough) of blood levels of p-tau-217, as measured by SIMOA blood neuro-metabolite assays.
Changes in sleep-wake amplitudes (peak-trough) of blood levels of glial fibrillary acidic protein (GFAP) | Pre- and 2 weeks post-intervention
  Difference between the CPAP on and CPAP off conditions in sleep-wake amplitudes (peak-trough) of blood levels of GFAP, as measured by SIMOA blood neuro-metabolite assays.
Changes in sleep-wake amplitudes (peak-trough) of blood levels of neurofilament light chain (NfL) | Pre- and 2 weeks post-intervention
  Difference between the CPAP on and CPAP off conditions in sleep-wake amplitudes (peak-trough) of blood levels of NfL, as measured by SIMOA blood neuro-metabolite assays.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Wong, MBBS FRACP, Principal Investigator — Woolcock Institute of Medical Research; Svetlana Postnova, PhD, Principal Investigator — University of Sydney; Mark Butlin, PhD, Principal Investigator — Macquarie University
Locations (1):
- Woolcock Institute of Medical Research, Macquarie Park, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holth JK, Fritschi SK, Wang C, Pedersen NP, Cirrito JR, Mahan TE, Finn MB, Manis M, Geerling JC, Fuller PM, Lucey BP, Holtzman DM. The sleep-wake cycle regulates brain interstitial fluid tau in mice and CSF tau in humans. Science. 2019 Feb 22;363(6429):880-884. doi: 10.1126/science.aav2546. Epub 2019 Jan 24. PMID 30679382
- [Background] Kang JE, Lim MM, Bateman RJ, Lee JJ, Smyth LP, Cirrito JR, Fujiki N, Nishino S, Holtzman DM. Amyloid-beta dynamics are regulated by orexin and the sleep-wake cycle. Science. 2009 Nov 13;326(5955):1005-7. doi: 10.1126/science.1180962. Epub 2009 Sep 24. PMID 19779148
- [Background] Bubu OM, Andrade AG, Umasabor-Bubu OQ, Hogan MM, Turner AD, de Leon MJ, Ogedegbe G, Ayappa I, Jean-Louis G G, Jackson ML, Varga AW, Osorio RS. Obstructive sleep apnea, cognition and Alzheimer's disease: A systematic review integrating three decades of multidisciplinary research. Sleep Med Rev. 2020 Apr;50:101250. doi: 10.1016/j.smrv.2019.101250. Epub 2019 Dec 12. PMID 31881487
- [Background] Iliff JJ, Wang M, Liao Y, Plogg BA, Peng W, Gundersen GA, Benveniste H, Vates GE, Deane R, Goldman SA, Nagelhus EA, Nedergaard M. A paravascular pathway facilitates CSF flow through the brain parenchyma and the clearance of interstitial solutes, including amyloid beta. Sci Transl Med. 2012 Aug 15;4(147):147ra111. doi: 10.1126/scitranslmed.3003748. PMID 22896675
- [Background] Xie L, Kang H, Xu Q, Chen MJ, Liao Y, Thiyagarajan M, O'Donnell J, Christensen DJ, Nicholson C, Iliff JJ, Takano T, Deane R, Nedergaard M. Sleep drives metabolite clearance from the adult brain. Science. 2013 Oct 18;342(6156):373-7. doi: 10.1126/science.1241224. PMID 24136970
- [Background] Bucks RS, Olaithe M, Rosenzweig I, Morrell MJ. Reviewing the relationship between OSA and cognition: Where do we go from here? Respirology. 2017 Oct;22(7):1253-1261. doi: 10.1111/resp.13140. Epub 2017 Aug 4. PMID 28779504
- [Background] Leng Y, McEvoy CT, Allen IE, Yaffe K. Association of Sleep-Disordered Breathing With Cognitive Function and Risk of Cognitive Impairment: A Systematic Review and Meta-analysis. JAMA Neurol. 2017 Oct 1;74(10):1237-1245. doi: 10.1001/jamaneurol.2017.2180. PMID 28846764
- [Background] Yaffe K, Laffan AM, Harrison SL, Redline S, Spira AP, Ensrud KE, Ancoli-Israel S, Stone KL. Sleep-disordered breathing, hypoxia, and risk of mild cognitive impairment and dementia in older women. JAMA. 2011 Aug 10;306(6):613-9. doi: 10.1001/jama.2011.1115. PMID 21828324
- [Background] Ju YS, Zangrilli MA, Finn MB, Fagan AM, Holtzman DM. Obstructive sleep apnea treatment, slow wave activity, and amyloid-beta. Ann Neurol. 2019 Feb;85(2):291-295. doi: 10.1002/ana.25408. Epub 2019 Jan 17. PMID 30597615